CLINICAL TRIAL: NCT00928564
Title: Addition of Pudendal Blocks to Pelvic Floor Physical Therapy for the Treatment of Pelvic Floor Tension Myalgia: A Randomized Controlled Trial
Brief Title: Addition of Pudendal Blocks to Pelvic Floor Physical Therapy for the Treatment of Pelvic Floor Tension Myalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Felicia Lane, Associate Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2009-6784
Record Dates: First submitted 2009-06-24; First posted 2009-06-26 (Estimated); Results first posted 2021-02-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-01

CONDITIONS: Pelvic Floor Muscle Spasm
Keywords: Pelvic floor muscle spasm; Pelvic pain; physical therapy; pudendal block
MeSH Terms: conditions — Pelvic Pain | interventions — Pharmaceutical Preparations; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pudendal Block (Active Comparator): 8ml of 0.5% bupivicaine, 1ml of 10mg/ml triamcinolone, 1ml of 8.4% sodium bicarbonate for a total volume of 10ml. Five ml will be used at each block site.
  Interventions: Drug: Pudendal block
- Placebo (Placebo Comparator): 5ml of saline at each block site
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pudendal block — 8ml of 0.5% bupivicaine, 1ml of 10mg/ml triamcinolone, 1ml of 8.4% sodium bicarbonate for a total volume of 10ml. Five ml will be used at each block site.
  Other Names: regional nerve block anesthesia (drug)
  Arms: Pudendal Block
Drug: Placebo — 5ml of saline at each block site.
  Other Names: saline
  Arms: Placebo

SUMMARY:
Pelvic floor tension myalgia (PFTM) is increasingly noted in patients with chronic pelvic pain. Pelvic floor physical therapy is typically utilized and is at times combined with other therapies such as botox injections, trigger point injections or pudendal blocks. The investigators' study will randomize newly diagnosed patients with PFTM to weekly . Final patient assessment will be performed at 6 months to assess durability of response.

Primary hypothesis: The addition of pudendal blocks to standard pelvic floor physical therapy will result in lower pain and pelvic floor muscle tension scores, lower baseline vaginal pressure and increase pelvic floor strength.

Secondary hypothesis: The addition of pudendal blocks to standard pelvic floor physical therapy will result in a lower pain score in a shorter time frame, resulting in faster progress through physical therapy.

DETAILED DESCRIPTION:
Participants will be identified within UC Irvine urogynecology and/or pelvic floor physical therapy practice with the underlying diagnosis of pelvic floor tension myalgia. This diagnosis may be secondary to various underlying etiologies including interstitial cystitis/painful bladder syndrome, vulvodynia, endometriosis, adhesive disease, unknown etiology, etc. At the time of enrollment, participants will be randomized into one of two groups: either standard pelvic floor physical therapy with weekly saline placebo injections or standard pelvic floor physical therapy and weekly pudendal blocks for 6 weeks. Standard physical therapy techniques will be utilized in both groups. Weekly injections of a mixture of a steroid and local anesthetic or saline will be administered depending on the randomization. Injections will be administered by a urogynecology physician. The participant and the treating physical therapist will be blinded to treatment assignment. The participant will be evaluated with for pelvic floor muscle strength and tenderness and will have pain assessed by a visual analog scale at baseline, weekly throughout the study, and at 6 months after study enrollment. Vaginal electromyography will be performed and standardized questionnaires regarding pelvic floor symptoms, quality of life and sexual function will be administered at baseline, after 6 weeks of injections and at 6 months after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant women over the age of 18 with the diagnosis of pelvic floor tension myalgia that are naive to pelvic floor physical therapy.
* Able to provide informed consent.
* Subjects must be willing to accept randomization.

Exclusion Criteria:

* Previously treated with physical therapy.
* An allergy to any component within the pudendal block.
* Bleeding disorders.
* Active vaginal infection.
* Inability to complete the questionnaires.
* Inability to read English (validated questionnaires are available in English only).
* Inability to complete the follow-up visits.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-04; Primary Completion 2015-12 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Felicia Lane, MD, Principal Investigator — University of California, Irvine
Locations (1):
- UCI Women's Healthcare, Orange, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pudendal Block | Placebo
Started | 28 | 12
Completed | 22 | 12
Not Completed | 6 | 0
Not completed — Lost to Follow-up | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pudendal Block | Placebo | Total
Number analyzed (Participants) | 28 | 12 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 12 | 40
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (3) | 45 (4) | 46 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 12 | 40
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 23 | 10 | 33
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 28 | 12 | 40

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Pain Score After 6 Weekly Injections
Description: 10 point likert scale to report pain a score from zero for no pain to ten for the worst possible pain
Time Frame: up to 8 weeks
Measure: Mean (Standard Deviation); unit: Visual Analog Pain Score
Arm/Group | Pudendal Block | Placebo
Number analyzed (Participants) | 22 | 12
Visual Analog Pain Score | 3.33 (1.87) | 2.99 (2.03)

2. Secondary Outcome: Improvement in Pelvic Floor Symptoms as Assessed Through Validated Questionnaires
Description: The Pelvic Floor Distress Inventory (PFDI) has 20 items and 3 scales, the response scale is from 0-4. Summary scores range from 0-300 with higher scores indicating more distress.
Time Frame: up to 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pudendal Block | Placebo
Number analyzed (Participants) | 22 | 12
score on a scale | 47.2 (30.8) | 38.2 (29)

ADVERSE EVENTS:
Time Frame: 6 weeks post treatment.
Arm/Group | Pudendal Block | Placebo
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/12
Other Adverse Events (participants affected / at risk) | 4/22 | 4/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pudendal Block (N=22) | Placebo (N=12)
vaginal bleeding (Surgical and medical procedures) | 2 | 4 — Eight Dindo grade one complications occurred during the study period. 6 vaginal bleeding, 2 toe numbness
Toe numbness (Surgical and medical procedures) | 2 | 0 — Transient toe numbness.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No